CLINICAL TRIAL: NCT01119456
Title: Phase 1 Study of the Anti-Ron Receptor Monoclonal Antibody IMC-RON8 in Patients With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or for Whom No Standard Therapy is Available
Brief Title: A Study of IMC-RON8 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 13958; CP21-0901 (Other: ImClone Systems); I5D-IE-JRCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Cancer
Keywords: Tumors; Macrophage stimulating 1 receptor, human; RON protein; RON receptor protein tyrosine kinase
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-RON8 (Experimental): A monoclonal antibody to human macrophage-stimulating 1-receptor-8 (RON8).
  Interventions: Biological: IMC-RON8

INTERVENTIONS:
Biological: IMC-RON8 — 5 milligrams per kilogram (mg/kg) intravenously (IV)
  Once a week for each 4-week treatment cycle, for a total of four doses per cycle. The initial 4-week treatment cycle will be followed by a 2-week observation period.
  Cohort 1
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 10 mg/kg IV
  Once a week for each 4-week treatment cycle, for a total of four doses per cycle. The initial 4-week treatment cycle will be followed by a 2-week observation period.
  Cohort 2
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 15 mg/kg IV
  Once a week for each 4-week treatment cycle, for a total of four doses per cycle. The initial 4-week treatment cycle will be followed by a 2-week observation period.
  Cohort 3
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 15 mg/kg IV
  Once every 2 weeks for each 4-week treatment cycle, for a total of two doses per cycle.
  Cohort 4
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 20 mg/kg IV
  Once every 2 weeks for each 4-week treatment cycle, for a total of two doses per cycle.
  Cohort 5
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 25 or 30 mg/kg IV
  Once every 2 weeks for each 4-week treatment cycle, for a total of two doses per cycle.
  Cohort 6
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 30, 35, or 40 mg/kg IV
  Once every 2 weeks for each 4-week treatment cycle, for a total of two doses per cycle.
  Cohort 7
  Other Names: Narnatumab; LY3012219
Biological: IMC-RON8 — 20 or 25 mg/kg IV
  Once every week for each 4-week treatment cycle, for a total of four doses per cycle.
  Cohort 8
  Other Names: Narnatumab; LY3012219

SUMMARY:
A dose escalation study to determine the maximum tolerated dose of IMC-RON8 in participants with solid tumors. Participants can either be dosed once a week, or once every other week.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically-confirmed advanced primary or recurrent solid tumors that have not responded to standard therapy or for which no standard therapy is available
* The participant has measurable or non-measurable disease
* The participant has not received major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy within 28 days prior to the first dose of study therapy
* The participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2
* The participant has adequate hematologic function
* The participant has adequate renal function as defined by serum creatinine ≤1.5 times the institutional upper limit of normal (ULN)
* The participant has a life expectancy >3 months

Exclusion Criteria:

* The participant has received chemotherapy or therapeutic radiation therapy within 28 days prior to the first dose of study therapy
* The participant has ongoing toxicities of >Grade 1 associated with any prior treatment
* The participant has a known sensitivity to monoclonal antibodies or other therapeutic agents, or to agents of similar biologic composition as IMC-RON8
* The participant has received treatment with any monoclonal antibodies within 6 weeks prior to first dose of study therapy
* The participant has received treatment with agents specifically targeting the RON ligand or receptor within 6 weeks prior to first dose of study therapy
* The participant has undergone a major surgical procedure, open biopsy, or experienced a significant traumatic injury within 28 days prior to the first dose of study therapy
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia (well controlled atrial fibrillation is permitted), psychiatric illness/social situations, active bleeding, or any other serious uncontrolled medical disorders in the opinion of the investigator
* The participant has known or suspected brain or leptomeningeal metastases (participants with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and may not be taking steroids; participants receiving anticonvulsants are eligible)
* The participant has a serious or nonhealing active wound, ulcer, or bone fracture
* The participant is currently using or has received a thrombolytic agent within 28 days prior to first dose of study therapy
* The participant is receiving full-dose warfarin (participants receiving low-dose warfarin to maintain the patency of permanent, indwelling intravenous catheters are eligible if the international normalized ratio is <1.5)
* The participant is receiving intravenous heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this dose escalation study, a completed participant was either a participant who completed the initial 4-week treatment cycle (and 2-weeks of observation for specified treatment arms) or one who discontinued therapy, during the same time period, for a narnatumab (IMC-RON8)-related toxicity.
Groups:
- IMC-RON8 (5 mg/kg qw): IMC-RON8: 5 mg/kg IMC-RON8 administered IV qw for a total of 4 doses per cycle. The initial 4-week treatment cycle was followed by a 2-week observation period. Following the first 6-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- IMC-RON8 (10 mg/kg qw): IMC-RON8: 10 mg/kg IMC-RON8 administered IV qw for a total of 4 doses per cycle.
  The initial 4-week treatment cycle was followed by a 2-week observation period. Following the first 6-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- IMC-RON8 (15 mg/kg qw): IMC-RON8: 15 mg/kg IMC-RON8 administered IV qw for a total of 4 doses per cycle.
  The initial 4-week treatment cycle was followed by a 2-week observation period. Following the first 6-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- IMC-RON8 (20 mg/kg qw): IMC-RON8: 20 mg/kg IMC-RON8 administered IV qw for a total of 4 doses per cycle.
  Participants continued treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met
- IMC-RON8 (15 mg/kg q2w): IMC-RON8: 15 mg/kg IMC-RON8 administered IV q2w for a total of 2 doses per cycle.
  Following the first 8-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met
- IMC-RON8 (20 mg/kg q2w): IMC-RON8: 20 mg/kg IMC-RON8 administered IV q2w for a total of 2 doses per cycle.
  Following the first 8-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- IMC-RON8 (30 mg/kg q2w): IMC-RON8: 30 mg/kg IMC-RON8 administered IV q2w for a total of 2 doses per cycle.
  Following the first 8-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- IMC-RON8 (40 mg/kg q2w): IMC-RON8: 40 mg/kg IMC-RON8 administered IV q2w for a total of 2 doses per cycle.
  Following the first 8-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Started | 7 | 3 | 3 | 13 | 4 | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 7 | 3 | 3 | 13 | 4 | 3 | 3 | 3
Completed | 7 | 3 | 3 | 13 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Participants who received at least 1 dose of study drug.
Groups:
- IMC-RON8 (20 mg/kg q2w: IMC-RON8: 20 mg/kg IMC-RON8 administered IV q2w for a total of 2 doses per cycle.
  Following the first 8-week tumor assessment, participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w) | IMC-RON8 (20 mg/kg qw) | Total
Number analyzed (Participants) | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (17.2) | 66.0 (2.0) | 65.3 (9.8) | 70.5 (9.1) | 57.7 (9.1) | 38.0 (13.1) | 67.3 (6.0) | 58.7 (11.6) | 59.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 1 | 4 | 1 | 2 | 1 | 3 | 17
  Male | 2 | 3 | 2 | 0 | 2 | 1 | 2 | 10 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4
  White | 7 | 3 | 3 | 3 | 3 | 3 | 2 | 9 | 33
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of IMC-RON8
Description: The MTD was the previous dose level to that in which 2 of 6 participants experienced dose-limiting toxicities (DLTs). DLTs were defined as any of the following events: Grade 4 neutropenia lasting >7 days; any Grade 3 or 4 neutropenia complicated by fever ≥38.5 degrees Celsius or infection, Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia complicated by hemorrhage; Grade 3 hepatic toxicity; or any Grade 3 or 4 nonhematologic toxicity (excluding alopecia, fatigue, anorexia, nausea, and vomiting that is controlled with antiemetics).
Time Frame: Baseline through end of study treatment (up to 48 weeks)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- IMC-RON8: IMC-RON8: Escalating doses (up to 40 mg/kg IMC-RON8) administered IV either qw or q2w for each 4-week cycle.
  Participants who responded to treatment (CR, PR, or SD) could continue treatment (same dose and frequency with no rest period) until PD, toxicity, or other withdrawal criteria were met.
Arm/Group | IMC-RON8
Number analyzed (Participants) | 39
mg/kg | NA — Because only 1 DLT was observed in the study, data were insufficient to determine the MTD.

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of IMC-RON8
Description: The Cmax of IMC-RON8 following the first and multiple IV infusions (the fourth infusion for the qw treatment regimen and the fifth infusion for the q2w treatment regimen) is reported. PK samples were collected per protocol and individual sampling times varied depending on the treatment arm and infusion (first or multiple). The geometric mean and geometric coefficient of variation (%CV) were calculated for treatment arms that had ≥3 participants who had evaluable PK samples for Cmax.
Time Frame: First and fourth or fifth infusion: Predose, immediately postdose through 168 or 336 hours postdose
Population: Participants who received a first and/or fourth or fifth dose of study drug and had evaluable PK samples for Cmax. No participant was analyzed for the geometric mean (%CV) of Cmax after multiple infusions in the 15, 20, 30, and 40 q2w treatment arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Number analyzed (Participants) | 7 | 3 | 3 | 13 | 4 | 3 | 3 | 3
micrograms per milliliter (mcg/mL)
  First infusion | 111 (31) | 183 (24) | 369 (20) | 437 (20) | 379 (17) | 506 (39) | 581 (7) | 706 (24)
  Multiple infusions: number analyzed (Participants) | 5 | 3 | 3 | 9 | 1 | 0 | 0 | 2
  Multiple infusions | 139 (50) | 263 (17) | 452 (29) | 518 (25) | NA (NA) — <3 participants. The participants individual value is 560.97. |  |  | NA (NA) — <3 participants. The participants individual values were 1055.57 and 711.99.

3. Secondary Outcome: PK: Area Under the Curve (AUC) of IMC-RON8
Description: The AUC from time 0 to the last quantifiable concentration [AUC(0-tlast)] of IMC-RON8 following the first IV infusion is reported along with the AUC for 1 dosing interval (AUC tau). Tau = fourth infusion through 168 hours post infusion for the qw regimen and the fifth infusion through 336 hours post infusion for the q2w regimen. PK samples were collected per protocol and individual sampling times varied depending on the treatment arm and infusion (first or multiple). The geometric mean and geometric coefficient of variation (%CV) were calculated for treatment arms that had ≥3 participants who had evaluable PK samples for AUC(0-tlast) or AUC tau.
Time Frame: First and fourth or fifth infusion: Predose, immediately postdose through 168 or 336 hours postdose
Population: Participants who received a first and/or fourth or fifth dose of study drug and had evaluable PK samples for AUC(0-tlast) or AUC tau. No participant was analyzed for the geometric mean (%CV) of AUC tau in the 15, 20, 30, and 40 q2w treatment arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (mcg*h/mL)
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Number analyzed (Participants) | 5 | 3 | 3 | 12 | 4 | 3 | 3 | 3
micrograms*hour/milliliter (mcg*h/mL)
  AUC(0-tlast): number analyzed (Participants) | 4 | 3 | 3 | 12 | 4 | 3 | 3 | 3
  AUC(0-tlast) | 8320 (63) | 12500 (14) | 23800 (37) | 29000 (30) | 35600 (22) | 40500 (87) | 56900 (34) | 70200 (25)
  AUC tau: number analyzed (Participants) | 5 | 3 | 3 | 6 | 1 | 0 | 0 | 2
  AUC tau | 10400 (87) | 19400 (11) | 31500 (51) | 29900 (47) | NA (NA) — n <3 participants. The participants individual value was 560.97. |  |  | NA (NA) — n <3 participants. The participants individual values were 113000 and 72200.

4. Secondary Outcome: Immunogenicity of IMC-RON8
Description: An immunogenicity assay for IMC-RON8 was not developed due to the decision to not further develop IMC-RON8 based on preliminary results of this study.
Time Frame: Prior to first infusion through study completion (up to 52 weeks)
Population: Zero participants analyzed. Immunogenicity data were not collected.
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Pharmacodynamics: H-Score of Macrophage-Stimulating 1-Receptor-8 (RON8)
Description: The expression of RON8 was measured in cell membrane/cytoplasm by immunohistochemistry (IHC) methods that incorporated both intensity and distribution of staining. The H-Score was calculated by summing the percentage of cell staining at each intensity multiplied by the weighted intensity of staining: 0 (no staining), 1+ (weak staining), 2+ (medium staining), 3+ (strongest staining). H-Scores could range from a minimum score of 0 to a maximum score of 300; the maximum score indicated the strongest expression. Pharmacodynamic samples were collected per protocol and individual sampling times varied depending on the treatment group.
Time Frame: Prior to first infusion through 1 hour post last infusion (end of study treatment, up to 48 weeks)
Population: Participants who received at least 1 dose of study drug and had tumor tissue samples.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w) | IMC-RON8 (20 mg/kg qw)
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 4 | 3 | 11
units on a scale | 80 [50 to 125] | 45 [0 to 90] | 60 [0 to 120] | 95 [50 to 140] | 133 [40 to 160] | 40 [0 to 120] | 40 [20 to 94] | 120 [0 to 200]

6. Secondary Outcome: Best Overall Tumor Response (Antitumor Activity of IMC-RON8 in the Treatment of Solid Tumors)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST, v 1.1) criteria. CR was the disappearance of all target and nontarget lesions; and any pathological lymph node (whether target or nontarget) must have had a reduction in short axis to <10 millimeters (mm) and normalization of tumor marker level of nontarget lesions. The disappearance of any intratumoral arterial enhancement in all target lesions was also required. PR was having at least a 30% decrease in sum of longest diameter of target lesions. PD was having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir and the unequivocal progression of existing nontarget lesions. SD was small changes that did not meet the above criteria.
Time Frame: Baseline to measured PD (up to 48 weeks)
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w) | IMC-RON8 (20 mg/kg qw)
Number analyzed (Participants) | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 13
Participants
  SD | 1 | 2 | 0 | 3 | 0 | 1 | 2 | 2
  PD | 4 | 1 | 3 | 0 | 2 | 2 | 1 | 8
  Unknown | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 3

7. Other Pre Specified Outcome: Number of Participants Who Died
Description: The number of participants who died is reported by cause of death.
Time Frame: Baseline through study completion (up to 52 weeks)
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Number analyzed (Participants) | 7 | 3 | 3 | 13 | 4 | 3 | 3 | 3
Participants
  Death Due to PD | 3 | 1 | 1 | 4 | 1 | 1 | 0 | 0
  Death, Cause Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | IMC-RON8 (5 mg/kg qw) | IMC-RON8 (10 mg/kg qw) | IMC-RON8 (15 mg/kg qw) | IMC-RON8 (20 mg/kg qw) | IMC-RON8 (15 mg/kg q2w) | IMC-RON8 (20 mg/kg q2w) | IMC-RON8 (30 mg/kg q2w) | IMC-RON8 (40 mg/kg q2w)
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/3 | 0/3 | 6/13 | 2/4 | 2/3 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 6/7 | 3/3 | 3/3 | 11/13 | 4/4 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-RON8 (5 mg/kg qw) (N=7) | IMC-RON8 (10 mg/kg qw) (N=3) | IMC-RON8 (15 mg/kg qw) (N=3) | IMC-RON8 (20 mg/kg qw) (N=13) | IMC-RON8 (15 mg/kg q2w) (N=4) | IMC-RON8 (20 mg/kg q2w) (N=3) | IMC-RON8 (30 mg/kg q2w) (N=3) | IMC-RON8 (40 mg/kg q2w) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IMC-RON8 (5 mg/kg qw) (N=7) | IMC-RON8 (10 mg/kg qw) (N=3) | IMC-RON8 (15 mg/kg qw) (N=3) | IMC-RON8 (20 mg/kg qw) (N=13) | IMC-RON8 (15 mg/kg q2w) (N=4) | IMC-RON8 (20 mg/kg q2w) (N=3) | IMC-RON8 (30 mg/kg q2w) (N=3) | IMC-RON8 (40 mg/kg q2w) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 2 (3) | 2 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (2) | 1 (2) | 2 (4) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (2) | 0 (0) | 7 (12) | 3 (8) | 1 (1) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile output abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (9) | 2 (3) | 2 (2) | 2 (3) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/2 (0) | 0 (0) | 1/2 (1) | 0/10 (0) | 0/0 (0) | 0/2 (0) | 0/1 (0) | 0/2 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/5 (0) | 0/0 (0) | 0/1 (0) | 0/3 (0) | 0 (0) | 0/1 (0) | 1/2 (1) | 0/1 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.